CLINICAL TRIAL: NCT06180317
Title: The Effect of Virtual Reality on Anxiety and Pain During Endometrial Biopsy: A Randomised Controlled Experimental Study
Brief Title: The Effect of Virtual Reality on Anxiety and Pain During Endometrial Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Associate Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KırklareliED-3
Record Dates: First submitted 2023-12-11; First posted 2023-12-22 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Endometrial Biopsy
Keywords: Endometrial Biopsy; Virtual Reality; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Experimental): Virtual reality to be applied to women undergoing endometrial biopsy.
  Interventions: Other: Virtual reality
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practive on their own to reduce anxiety and pain during endometrial biopsy.

INTERVENTIONS:
Other: Virtual reality — Participants will view a specific relaxing and distracting scenario using virtual reality (VR) for approximately 7-8 minutes from one minute before the procedure until the end of the procedure. Assessment will be performed with STAI and VAS just before the endometrial biopsy procedure, VAS during the procedure and again with STAI and VAS after the procedure.
  Arms: Virtual reality group

SUMMARY:
The aim of this study was to reduce the anxiety and pain felt during endometrial biopsy procedure.

DETAILED DESCRIPTION:
Endometrial cancers are among the most common gynaecological cancers globally, while abnormal uterine bleeding is a common gynaecological problem.Endometrial biopsy is a safe method frequently used in gynaecology to evaluate abnormal or postmenopausal uterine bleeding. It is a rapid and cost-effective medical procedure performed to examine the endometrium to detect the presence of endometrial hyperplasia, malignancy or other pathological conditions.

Since early diagnosis and correct treatment can affect the prognosis of the disease, endometrial biopsy is considered an important diagnostic and screening tool for women's health. Although endometrial biopsy is a painless or mildly painful procedure, approximately half of the patients experience pain of different intensity during the procedure.Endometrial biopsy, which is an invasive procedure, can trigger anxiety in women and increase the perceived pain experience and severity by reducing pain tolerance during the procedure.

Effective management of anxiety, which can also exacerbate the pain experienced during endometrial biopsy procedure, can increase women's comfort and satisfaction. Therefore, anxiety management may be effective in helping women cope with the problems experienced during the endometrial biopsy procedure. While many alternative methods are used to reduce anxiety in the literature (acupressure, meditation, laughter therapy, art therapy), the therapeutic effect of virtual reality has also been reported in studies.

Virtual reality (VR) is an interactive virtual environment dating back to the 1960s, where the user experiences the virtual world by feeling "there" in the virtual world thanks to computer technologies. It represents complex technologies in which visual, auditory and tactile multisensory inputs are integrated into a 3D environment. It is a virtual space that can include hand or body tracking sensors with a VR headset and expands up to 360 degrees, offering users experiences similar to those in the real world. In addition, VR is frequently used in various sectors such as education, gaming, simulation and design, as well as in the field of health. A randomised clinical trial by Chiu et al. showed that virtual reality was effective in reducing anxiety in patients. The results of another study conducted by Yamashita et al. revealed that virtual reality improved anxiety and pain.

When the studies in the literature were examined, no study on the effect of virtual reality on anxiety and pain that may be experienced during endometrial biopsy procedure was found. In this study, it was aimed to determine the effect of virtual reality use on anxiety and pain during endometrial biopsy.

ELIGIBILITY:
Inclusion Criteria:

* -Volunteering to participate in the research
* Answering questionnaire and scale forms completely
* Ability to read and understand Turkish
* 18 years of age or older
* STAI score of 35 and above

Exclusion Criteria:

* Unwilling to continue working
* Having any problem that prevents communication (such as impaired hearing, speech, comprehension skills),
* Having used a pharmacological agent with analgesic or anxiolytic effect or a non-pharmacological method 24 hours before the procedure
* Having any psychiatric illness
* Vertigo, vision, hearing, perception problems
* Pregnancy
* Acute pelvic inflammatory disease, acute cervical and vaginal infection

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 80 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | between one to six months
  The form consists of questions about socio-demographic and endometrial biopsy

SECONDARY OUTCOMES:
The State/Trait Anxiety Inventory (STAI) | between one to six months
  This inventory was developed by Spielberg in 1973 and each of the subscales ranges from 1 (not at all) to 4 (very much). The lowest and highest scores that can be obtained from each subscale are 20 and 80, respectively. Higher scores are associated with more anxiety. The alpha value of the scale varies between 0.86 and 0.92 . Öner et al. 1983, it was shown that the alpha value of the Turkish version of the STAI ranged between 0.83 and 0.87.27.
Visual Anolag Scale (VAS) | between one to six months
  It was developed by Price et al. (1983) to assess the severity of pain. It is a line, usually 10 cm long, horizontal or vertical, starting with "No Pain" and ending with "Intolerable Pain". This line may be just a straight line, or it may be divided into equal intervals, or it may have description words placed on the line to describe pain. It is generally accepted that the vertical line is easier to understand. The patient indicates the intensity of his/her pain with a mark on this line where he/she deems appropriate. The distance between the beginning of no pain and this point is measured in "cm" and recorded. Values vary between 0 and 10 and higher values indicate increased pain. Turkish validity and reliability was performed by Eti Aslan.

CONTACTS AND LOCATIONS:
Overall Officials: meltem yavuz, Midwife, Principal Investigator — 1. Murat state hospital
Locations (1):
- 1.Murat State Hospital, Edirne, Turkey (Türkiye)